CLINICAL TRIAL: NCT01689077
Title: Time-differentiated Treatment With Mild Therapeutic Hypothermia Following Cardiac Arrest, a Multi Center Study.
Brief Title: Time-differentiated Therapeutic Hypothermia
Acronym: TTH48
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TTH48
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-12

CONDITIONS: Out of Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Hypothermia, Induced

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 24 hours hypothermia (Active Comparator): 24 hours hypothermia
  Interventions: Other: Therapeutic hypothermia
- 48 hours hypothermoa (Experimental): 48 hours hypothermia
  Interventions: Other: Therapeutic hypothermia

INTERVENTIONS:
Other: Therapeutic hypothermia — Mild therapeutic hypothermia with a target temperature of 33 degrees Centigrade for 24 or 48 hours

SUMMARY:
The purpose of this study is to determine if 48 hours of mild therapeutic hypothermia following out of hospital cardiac arrest gives a better cerebral outcome compared to 24 hours therapeutic hypothermia.

DETAILED DESCRIPTION:
Sudden out-of-hospital cardiac arrest (OOH-CA) remains a significant cause of death. However, in 2002 it was in two clinical trials demonstrated that mild therapeutic hypothermia in comatose OOH-CA victims yields a better cerebral outcome measured by Cerebral Performance Category Score (CPC) after 6 month. The optimal mild hypothermia treatment time is however not known. The two trials from 2002 apply the treatment for 12 and 24 hours respectively. In newborns with cerebral hypoxic damage the standard treatment time is 72 hours. It is therefore relevant to investigate the influence of the treatment time on the cerebral outcome in OOH-CA victims. In the present study cerebral outcome after mild therapeutic hypothermia (target temperature 33 degrees centigrade) in OOH-CA patients for 24 is compared to outcome after 48 hours of mild hypothermia. The main outcome parameter is mortality and CPC score measured 6 month after the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Out of hospital cardiac arrest of suspected cardiac origin
2. Return of spontaneous circulation (ROSC)
3. Glasgow Coma Score < 8
4. Estimated time interval from cardiac arrest to ROSC ≤ 60 min

Exclusion Criteria:

1. OOH-CA of suspected origin other than cardiac
2. In hospital Cardiac arrest
3. Terminal disease
4. Coagulation disorders
5. Unwitnessed asystolia
6. Time from cardiac arrest to start of hypothermia treatment > 240 min
7. GCS ≥ 8
8. Pregnancy
9. Persistent cardiogenic shock (Systolic blood pressure < 80 mmHg despite inotropic treatment and aortic balloon pump).
10. CPC 3-4 before cardiac arrest
11. Acute intra cerebral bleeding
12. Acute stroke
13. Acute coronary artery bypass grafting

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2013-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
CPC | 6 month
  CPC = Cerebral Performance Category Score. The primary outcome of the study is analyzed as the proportion of patients with good neurological outcome in the two groups, (CPC 1-2) at 6 months after CA.

SECONDARY OUTCOMES:
Adverse events | 10 days
  Adverse events are registered during the treatment and until discharge from primary hospital unit
CPC at discharge | 3 month
  CPC at discharge from primary hospital unit and after 28 days plus after 3 month
Mortality | 6 month
  CPC 5 at 6 month

OTHER OUTCOMES:
GCS | 28 days
  Glasgow Coma Score at day 4 and at discharge from primary hospital unit
GCS progression | 25 weeks
  Glasgow Coma Score throughout the observation period

CONTACTS AND LOCATIONS:
Overall Officials: Hans Kirkegaard, Professor, Principal Investigator — Department of Anaesthesia and Intensive care medicine, Aarhus University Hosptal, Brendstrupgaardsvej 8200 Aarhus, Denmark
Locations (10):
- Department of Intensive Care, Erasme Hospital, Brussels, Belgium
- Denmark (4):
  - Department of Anesthesiology and Intensive Care Medicine, Aarhus University Hospital, Aalborg, Aalborg
  - Department og Anesthesiologi and Intensive Care Medicine,, Aarhus
  - Department of Cardiology, Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Department of Anaesthesiology and Intensive Care Medicine, Odense University Hospital, Odense
- Anaesthesiology Clinic, North Estonia Medical Centre, Tallinn, Estonia
- Finland (2):
  - Division of Anaesthesiology and Intensive Care Medicine, Department of Surgery, Helsinki University Central Hospital, Helsinki
  - Hospital District of Southwest Finland), Kiinamyllynkatu, Turku
- Department of Internal Medicine, Nephrology and Intensive Care; Charité-Universitätsmedizin Berlin, Berlin, Germany
- Anesthesiology and Critical Care, Stavanger University Hospital, Stavanger, Norway

REFERENCES:
- [Derived] Evald L, Skrifvars MB, Virta JJ, Tiainen M, Laitio T, Leithner C, Soreide E, Hassager C, Rasmussen B, Grejs AM, Jeppesen AN, Kirkegaard H, Nielsen JF. Long-term functional outcome and quality of life 5-8 years after out of hospital cardiac arrest. Resuscitation. 2025 Oct;215:110672. doi: 10.1016/j.resuscitation.2025.110672. Epub 2025 Jun 9. PMID 40499675
- [Derived] Larsen AI, Grejs AM, Vistisen ST, Strand K, Skadberg O, Jeppesen AN, Duez CHV, Kirkegaard H, Soreide E. Kinetics of 2 different high-sensitive troponins during targeted temperature management in out-of-hospital cardiac arrest patients with acute myocardial infarction: a post hoc sub-study of a randomised clinical trial. BMC Cardiovasc Disord. 2022 Jul 30;22(1):342. doi: 10.1186/s12872-022-02778-4. PMID 35907787
- [Derived] Bach HM, Duez CHV, Jeppesen AN, Strand K, Soreide E, Kirkegaard H, Grejs AM. MR-proANP and NT-proBNP During Targeted Temperature Management Following Out-of-Hospital Cardiac Arrest: A Post hoc Analysis of the TTH48 Trial. Ther Hypothermia Temp Manag. 2022 Jun;12(2):82-89. doi: 10.1089/ther.2021.0012. Epub 2021 Aug 10. PMID 34375135
- [Derived] Hastbacka J, Kirkegaard H, Soreide E, Taccone FS, Rasmussen BS, Storm C, Kjaergaard J, Laitio T, Duez CHV, Jeppesen AN, Grejs AM, Skrifvars MB. Severe or critical hypotension during post cardiac arrest care is associated with factors available on admission - a post hoc analysis of the TTH48 trial. J Crit Care. 2021 Feb;61:186-190. doi: 10.1016/j.jcrc.2020.10.026. Epub 2020 Nov 2. PMID 33181415
- [Derived] Skrifvars MB, Soreide E, Sawyer KN, Taccone FS, Toome V, Storm C, Jeppesen A, Grejs A, Duez CHV, Tiainen M, Rasmussen BS, Laitio T, Hassager C, Kirkegaard H. Hypothermic to ischemic ratio and mortality in post-cardiac arrest patients. Acta Anaesthesiol Scand. 2020 Apr;64(4):546-555. doi: 10.1111/aas.13528. Epub 2019 Dec 26. PMID 31830304
- [Derived] Evald L, Bronnick K, Duez CHV, Grejs AM, Jeppesen AN, Soreide E, Kirkegaard H, Nielsen JF. Prolonged targeted temperature management reduces memory retrieval deficits six months post-cardiac arrest: A randomised controlled trial. Resuscitation. 2019 Jan;134:1-9. doi: 10.1016/j.resuscitation.2018.12.002. Epub 2018 Dec 17. PMID 30572070
- [Derived] Kirkegaard H, Soreide E, de Haas I, Pettila V, Taccone FS, Arus U, Storm C, Hassager C, Nielsen JF, Sorensen CA, Ilkjaer S, Jeppesen AN, Grejs AM, Duez CHV, Hjort J, Larsen AI, Toome V, Tiainen M, Hastbacka J, Laitio T, Skrifvars MB. Targeted Temperature Management for 48 vs 24 Hours and Neurologic Outcome After Out-of-Hospital Cardiac Arrest: A Randomized Clinical Trial. JAMA. 2017 Jul 25;318(4):341-350. doi: 10.1001/jama.2017.8978. PMID 28742911
- [Derived] Kirkegaard H, Pedersen AR, Pettila V, Hjort J, Rasmussen BS, de Haas I, Nielsen JF, Ilkjaer S, Kaltoft A, Jeppesen AN, Grejs AM, Duez CH, Larsen AI, Toome V, Arus U, Taccone FS, Storm C, Laitio T, Skrifvars MB, Soreide E. A statistical analysis protocol for the time-differentiated target temperature management after out-of-hospital cardiac arrest (TTH48) clinical trial. Scand J Trauma Resusc Emerg Med. 2016 Nov 28;24(1):138. doi: 10.1186/s13049-016-0334-0. PMID 27894327
- [Derived] Kirkegaard H, Rasmussen BS, de Haas I, Nielsen JF, Ilkjaer S, Kaltoft A, Jeppesen AN, Grejs A, Duez CH, Larsen AI, Pettila V, Toome V, Arus U, Taccone FS, Storm C, Skrifvars MB, Soreide E. Time-differentiated target temperature management after out-of-hospital cardiac arrest: a multicentre, randomised, parallel-group, assessor-blinded clinical trial (the TTH48 trial): study protocol for a randomised controlled trial. Trials. 2016 May 4;17(1):228. doi: 10.1186/s13063-016-1338-9. PMID 27142588